CLINICAL TRIAL: NCT05704244
Title: A Phase 3, Open Label Trial to Evaluate the Safety and Efficacy of FE 999326 Administered Intravesically to Japanese Subjects With High-grade, BCG Unresponsive, Non-muscle Invasive Bladder Cancer (NMIBC)
Brief Title: Safety and Efficacy of FE 999326 Administered Intravesically to Japanese Subjects With High-grade, BCG Unresponsive, Non-muscle Invasive Bladder Cancer (NMIBC)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000381
Record Dates: First submitted 2022-12-21; First posted 2023-01-30 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FE 999326 (Experimental)
  Interventions: Drug: FE 999326

INTERVENTIONS:
Drug: FE 999326 — 75 mL FE 999326 (3 x 10^11 vp/mL) of sterile suspension instilled once every 3 months into the bladder via a urinary catheter
  Other Names: nadofaragene firadenovec

SUMMARY:
To evaluate the safety and efficacy of FE 999326 in Japanese subjects with high-grade, BCG unresponsive NMIBC.

ELIGIBILITY:
Inclusion Criteria:

* Have at entry, confirmed by a pathology report:

  1. Carcinoma in situ (CIS) only
  2. Ta/T1 high-grade disease with concomitant CIS or
  3. Ta/T1 high-grade disease without concomitant CIS
* Subjects who did not respond to BCG treatment and have a persistent high-grade recurrence within 12 months after BCG was initiated, and those who despite an initial complete response to BCG, relapse with CIS within 12 months of their last intravesical treatment with BCG or relapse with high-grade Ta/T1 NMIBC within 6 months of their last intravesical treatment with BCG.
* Life expectancy >2 years, in the opinion of the investigator
* Eastern Cooperative Oncology Group (ECOG) status 2 or less
* Absence of concomitant upper tract urothelial carcinoma or urothelial carcinoma within the prostatic urethra
* Subjects with prostate cancer on active surveillance at low risk for progression, defined as prostate-specific antigen (PSA) <10 ng/dL

Exclusion Criteria:

* Current or previous evidence of muscle invasive (muscularis propria) or metastatic disease presented at the screening visit.
* Current systemic therapy for bladder cancer
* Current or prior investigational treatment for BCG unresponsive NMIBC or any other investigational drug within 1 month prior to screening
* Current or prior pelvic external beam radiotherapy within 5 years of entry
* Use of other adenovirus vector medications, including COVID-19 vaccines, within 2 weeks before and after instillation
* History of malignancy of other organ system within past 5 years, except treated basal cell carcinoma or squamous cell carcinoma of the skin and ≤pT2 upper tract urothelial carcinoma at least 24 months after nephroureterectomy.
* Subjects who cannot hold instillation for 1 hour
* Subjects who cannot tolerate intravesical dosing or intravesical surgical manipulation
* Intravesical therapy within 8 weeks prior to beginning trial treatment, with the exception of:

  * Cytotoxic agents when administered as a single instillation immediately following a TURBT procedure
  * Previous intravesical BCG therapy
* Systemic immunosuppressive therapy within 3 months prior to screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Whether or not a subject with CIS (with or without concomitant high-grade Ta or T1 papillary disease) responds to treatment, defined as complete response at any time after first administration of FE 999326 | At Month 12 assessment
  A subject with CIS (with or without concomitant high-grade Ta or T1 papillary disease) has achieved a complete response at an efficacy assessment if urine cytology is negative and there are no lesions on cystoscopy. If biopsy of the bladder is performed, this must be negative.

SECONDARY OUTCOMES:
Duration of complete response in subjects with CIS (with or without concomitant high-grade Ta or T1 papillary disease) who show a complete response at any time after first administration of FE 999326 | Up to 5 years
Whether or not a subject with high-grade Ta or T1 papillary disease (without concomitant CIS) responds to treatment, defined as absence of recurrence of high-grade disease | Up to 4 years
Duration of event-free survival in subjects with high-grade Ta or T1 papillary disease (without concomitant CIS) and in subjects with CIS (with or without papillary disease) | Up to 5 years
Incidence of cystectomy | Up to 4 years
Time to cystectomy | Up to 4 years
Overall survival | Up to 5 years
Concentration of FE 999326-specific DNA levels in urine | Up to day 1 of month 4 after start of treatment; and 3, 6, 9 and 12 months after last dose (up to 5 years after start of treatment)
Type, incidence, relatedness and severity of treatment emergent adverse events | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (24):
- Japan (24):
  - Ferring Investigational Site, Nagakute-shi, Aichi-ken
  - Ferring Investigational Site, Nagoya, Aichi-ken
  - Ferring Investigational Site, Narita-shi, Chiba
  - Ferring Investigational Site, Matsuyama, Ehime
  - Ferring Investigational Site, Fukuoka, Fukuoka
  - Ferring Investigational Site, Hiroshima, Hiroshima
  - Ferring Investigational Site, Hakodate-shi, Hokkaido
  - Ferring Investigational Site, Sapporo, Hokkaido
  - Ferring Investigational Site, Hitachi-shi, Ibaraki
  - Ferring Investigational Site, Tsukuba, Ibaraki
  - Ferring Investigational Site, Kawasaki-shi, Kanagawa
  - Ferring Investigational Site, Yokohama, Kanagawa
  - Ferring Investigational Site, Nankoku-shi, Kochi
  - Ferring Investigational Site, Tsu, Mie-ken
  - Ferring Investigational Site, Sendai, Miyagi
  - Ferring Investigational Site, Matsumoto-shi, Nagano
  - Ferring Investigational Site, Kashihara-shi, Nara
  - Ferring Investigational Site, Okayama, Okayama-ken
  - Ferring Investigational Site, Takatsuki-shi, Osaka
  - Ferring Investigational Site, Bunkyo-ku, Tokyo
  - Ferring Investigational Site, Minato-ku, Tokyo
  - Ferring Investigational Site, Mitaka-shi, Tokyo
  - Ferring Investigational Site, Toyama, Toyama
  - Ferring Investigational Site, Wakayama, Wakayama

IPD SHARING:
Plan to Share IPD: No